CLINICAL TRIAL: NCT00591136
Title: Dose-finding and Pharmacokinetic Trial of Orally Administered D-24851 to Patients With Solid Tumors
Brief Title: Phase I Study of Indibulin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL1001
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — indibulin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: indibulin

INTERVENTIONS:
Drug: indibulin — Dose escalation, daily dosing for 14 days every 3 weeks, for up to 4 months
  Other Names: ZIO-301

SUMMARY:
Dose-finding and pharmacokinetic trial of orally administered Indibulin to patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Male or female patient, >= 18 years of age.
* Histologically/cytologically proven solid malignant tumor, for which standard treatment of proven efficacy are not or no longer available.
* Performance status 0-2 ECOG/WHO.
* Life expectancy > 3 months.
* Able and willing to undergo blood sampling for pharmacokinetics.
* Written informed consent.

Exclusion Criteria

* Safety concerns:
* Any non-compensated or uncontrolled non-malignant condition, such as, symptomatic heart failure, active tuberculosis or any other chronic or active infection.
* History of allergic reaction to one of the ingredients of the trial medication.
* Clinically relevant abnormality in organ function as evidenced by any of the following pa¬ra¬meters:
* White blood cell count: < 3.0 x 109/l ANC: < 1.5 x 109/l
* Thrombocytes: < 100 x 109/l
* Hemoglobin < 6.0 mM
* Bilirubin (total): > 1.5 times upper limit of normal range
* ASAT, ALAT: > 2.5 times upper limit of normal range unless related to metastases in which case > 5 times upper normal limit is allowed
* Creatinine (serum) > 135 µmol/l (> 1.5 mg/100ml) OR
* Creatinine clearance: < 50 ml/min (calculated according to modified Cockcroft and Gault)
* Breast feeding, pregnancy or planned pregnancy. A reliable method of contraception must be used in men and in women of childbearing potential during the study and for 3 months after last study drug administration.
* Lack of suitability for the trial:
* Concomitant treatment with any other investigational drugs or exposure to another investigational agent within the last 4 weeks prior to study specific screening procedures (period should be extended if the patient has received any drug which is known to have de¬layed toxicity or prolonged half-life).
* Active peptic ulcer or any GI condition that could alter absorption or motility.
* Chronic use of H2-antagonists or proton pump inhibitors.
* Any other cancer treatment during the study or administered within the last 4 weeks (6 weeks for nitrosoureas, mitomycin C, high-dose carboplatin or extensive radiotherapy) before start of study treatment, except irradiation of non-target lesions for symptom relief and bi-phosphonate treatment of bone metastases.
* Clinically symptomatic brain metastases or leptomeningeal disease.
* Neurological or psychiatric disease or drug or alcohol abuse which would interfere with the patients proper completion of the protocol assignment.
* Administrative reasons:
* Anticipated non-availability for study visits/procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
toxicities | 4 months

SECONDARY OUTCOMES:
pharmacokinetics | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, Study Director — ZIOPHARM Oncology, Inc
Locations (2):
- Netherlands (2):
  - Amsterdam
  - Utrecht

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268